CLINICAL TRIAL: NCT00276237
Title: Review of Outcomes Following Pulmonary Valve Replacement for Congenital Heart Disease in Adults
Brief Title: Outcomes Following Pulmonary Valve Replacement in Adults
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Brian Kogon, Principal Investigator, Emory University
Other Study IDs: 0668-2005
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Heart Disease, Congenital; Pulmonary Valve Replacement
Keywords: Congenital Heart Disease; Pulmonary Valve Replacement
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
One of the most common residual lesions in adult survivors of pediatric cardiac surgery is pulmonary valve disease, particularly regurgitation.

Multiple studies have demonstrated that placement of a pulmonary valve in such patients, results in improved ventricular function and resolution of symptoms. However, the optimal prosthetic valve for use in the pulmonary position has not been defined. There are essentially three alternatives available: the stented bioprosthetic valve, stentless bioprosthetic "tube" grafts used to replace the entire right ventricular outflow tract and mechanical valves.

All three of these valve options have been used in adults with congenital heart disease at Emory Healthcare and at Children's Healthcare of Atlanta at Egleston.

The goal of this study is to evaluate and compare the indications and short and mid-term outcomes for these alternative therapies.

ELIGIBILITY:
Inclusion Criteria: Adult patients who have received a pulmonary valve replacement for congenital heart disease at Children's Healthcare of Atlanta at Egleston or are in the Emory Healthcare System between 1976 and 2004.

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-07; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Kirshbom, MD, Principal Investigator — Emory University Medical Center
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory Healthcare System, Atlanta, Georgia